CLINICAL TRIAL: NCT01064934
Title: Randomized Controlled Trial of Efficacy and Safety of Lipid Apheresis for the Prevention of Cardiovasc. Events in Patients With Progr. Cardiovasc. Disease, Lp(a)≥ 60 mg/dl and LDL-C <130 mg/dl on Maximally Tolerated Lipid-lowering Therapy
Brief Title: Randomized Controlled Trial of Lipid Apheresis in Patients With Elevated Lipoprotein(a)
Acronym: ELAILa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Heiner K. Berthold, Professor, and Elisabeth Steinhagen-Thiessen, Professor, Charite University Medicine Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELAILa-01
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2010-05

CONDITIONS: Hyperlipoproteinemia(a); Progressive Cardiovascular Disease
Keywords: coronary heart disease; cerebrovascular disease; peripheral arterial disease; atherosclerosis; hyperlipoproteinemia
MeSH Terms: conditions — Coronary Disease; Cerebrovascular Disorders; Peripheral Arterial Disease; Atherosclerosis; Hyperlipoproteinemias | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipid apheresis (Experimental): Lipid apheresis
  Interventions: Procedure: Lipid apheresis
- Standard care (Active Comparator): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Lipid apheresis — Weekly lipid apheresis procedure for lipoprotein(a) lowering
  Arms: Lipid apheresis
Other: Standard care — Standard care for maximum cardiovascular risk reduction (behavioural, exercise, nutrition, drugs, etc.)
  Arms: Standard care

SUMMARY:
Lipoprotein(a) [Lp(a)] is an independent risk factor for cardiovascular disease. Non-medical treatment measures (e.g. dietary therapy or weight loss) can hardly influence Lp(a) plasma concentrations. Drug therapy has only limited influence, e.g. treatment with niacin. Statins are usually without effect. Lipid apheresis is the only treatment known to lower elevated Lp(a) levels in a relevant way. In patients with pronounced elevation of Lp(a) and normal LDL cholesterol levels, who suffer from progressive cardiovascular disease, the treatment with lipid apheresis seems to be a last-resort treatment option. The current trial will evaluate the effectiveness of lipid apheresis on cardioavascular endpoints.

DETAILED DESCRIPTION:
Lipoprotein(a) [Lp(a)] is an independent risk factor for cardiovascular disease. Non-medical treatment measures (e.g. dietary therapy or weight loss) can hardly influence Lp(a) plasma concentrations. Drug therapy has only limited influence, e.g. treatment with niacin. Statins are usually without effect. Lipid apheresis is the only treatment known to lower elevated Lp(a) levels in a relevant way. In patients with pronounced elevation of Lp(a) and normal LDL cholesterol levels, who suffer from progressive cardiovascular disease, the treatment with lipid apheresis seems to be a last-resort treatment option. The current trial will evaluate the effectiveness of lipid apheresis on cardioavascular endpoints. The trial is a randomized multicenter trial in Germany. Patients will be randomized to the apheresis group or to the control group. All patients will receive maximal risk minimizing therapies. The apheresis group will receive in addition weekly lipid apheresis. The principal outcome parameter is a composite endpoint of non-fatal myocardial infarction, interventional therapeutic procedure (PCI, stenting), coronary bypass surgery (CABG), non-fatal ischemic cerebrovascular accident, hospitalization due to acute coronary syndrome (ACS), critical limb ischemia, peripheral arterial revascularization procedure; amputation, death from cardiovascular cause.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Male or female
* Written informed consent
* Lipoprotein(a) >=60 mg/dL
* Low-density lipoprotein cholesterol <130 mg/dL
* Progressive cardiovascular disease
* Positive recommendation by the Inclusion Committee

Exclusion Criteria:

* Current participation in a lipid apheresis program
* Previous participation in a lipid apheresis program
* Low-density lipoprotein cholesterol >=130 mg/dL under maximally tolerated (or necessary) drug treatment
* Triglyceride concentrations >=450 mg/dL
* Known homozygous familial hypercholesterolemia
* Known type III hyperlipoproteinemia
* Pregnancy, breast feeding
* History of malignant disease (with the exception of non-melanoma carcinomas of the skin and carcinoma in situ of the cervix)
* Planned major surgical procedures in the next 3 months
* Current participation in another interventional trial
* Previous randomization in the current trial (applies only for the RCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint, defined as first occurrence of one of the following: myocardial infarction, interventional therapeutic procedure, CABG, cerebrovascular accident, hospitalization due to ACS, periph. art. revasc., death from cardiovascular cause | 5 years

SECONDARY OUTCOMES:
Components of the primary endpoint considered individually | 5 years
Death from any cause | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heiner K. Berthold, MD, PhD, Principal Investigator — Charite University, Berlin, Germany; Elisabeth Steinhagen-Thiessen, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Lipidambulanz, Interdisziplinäres Stoffwechsel-Centrum, CVK, Charite, Berlin, Germany